CLINICAL TRIAL: NCT06796725
Title: Prospective Exploratory Study on rTMS for Migraine Under the Guidance of MEG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Migraine-MEG-2024
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Migraine Disorders, Brain; rTMS Stimulation
Keywords: Migraine; MEG; rTMS; RCT
MeSH Terms: conditions — Migraine Disorders | interventions — Flunarizine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This study adopted a single blind approach, with evaluators being blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RTMS intervention group (Experimental): (1) The patient undergoes pseudo stimulus intervention in the first week and real stimulus intervention afterwards, which is blind to the patient. (2) Starting from the second week, true stimulation intervention will be conducted for 4 weeks, with each patient making an appointment for 1 month.
  Interventions: Device: rTMS
- Sibelium treatment group (Other): Patients were evaluated and followed up with a scale based on medication intervention.
  Interventions: Drug: Sibelium

INTERVENTIONS:
Device: rTMS — (1) The patient undergoes pseudo stimulus intervention in the first week and real stimulus intervention afterwards, which is blind to the patient. (2) Starting from the second week, true stimulation intervention will be conducted for 4 weeks, with each patient making an appointment for 1 month. On Day 7 after the patient intervention, Day 14, Day 30, Day 60, Day 90, Day 180 scales were used to evaluate follow-up.
  Arms: RTMS intervention group
Drug: Sibelium — Sibelium 10mg is taken orally every night for 4 weeks each course of treatment. Patients were evaluated and followed up with a scale based on medication intervention, including Day 7, Day 14, Day 30, Day 60, Day 90, and Day 180
  Arms: Sibelium treatment group

SUMMARY:
Using magnetoencephalography to locate and regulate targets in migraine patients, repeating transcranial magnetic stimulation to physically regulate targets, and evaluating the safety and effectiveness of this treatment method through headache related scales. Using whole genome data and scale scores for correlation analysis, and conducting randomized controls with traditional drugs to explore new approaches for migraine.

DETAILED DESCRIPTION:
Migraine patients who meet the inclusion criteria will be randomly divided into two groups: the MEG+rTMS treatment group and the Sibelium treatment group. Evaluate the clinical efficacy (frequency of attacks (times/month), severity (visual analog scale), duration (d), analgesic drug use rate, and related scale scores) of the MEG+rTMS treatment group and the Sibelium treatment group, respectively. Evaluate its efficacy based on follow-up results and analyze the correlation between different genotypes and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Complies with specific disease diagnosis: A. Headaches that meet the criteria of B and C (headaches that meet the characteristics of tension headaches or migraines) should occur at least 15 days per month and last for at least 3 months; B. Headaches that meet the criteria of 1.1 migraine without aura diagnosis B-D or 1.2 migraine with aura B and C occurring at least 5 times; C. Headache meets any of the following criteria and occurs for more than 8 days per month, lasting for more than 3 months: ①1.1 C and D of migraine without aura②1.2 B and C of migraine with aura③ The migraine attack perceived by the patient can be relieved by taking triptan or ergot, which cannot be better explained by other diagnoses in ICHD-3.
* Must be able to swallow tablets
* Signed and dated informed consent form Promise to comply with research procedures and cooperate in implementing the entire research process

Exclusion Criteria:

* Age under 15 years old; Accompanied by optic disc edema, focal symptoms and signs of the nervous system (except for typical visual and sensory precursors) or cognitive impairment; Sudden and rapidly peaking severe headaches (thunderous headaches)
* Accompanied by fever; New onset headaches in adults, especially after the age of 50; Headaches in patients with high coagulation risk
* New headache in patients with tumor or AIDS history; Headaches related to changes in body position;
* History of epileptic seizures

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Headache Scale Reduction Rate | From enrolment to the end of the 4-week treatment.
  Deduction rate=(score of therapeutic efficacy scale at different time points after treatment - score of therapeutic efficacy scale before treatment)/score of therapeutic efficacy scale before treatment. If the headache scale score decreases by 20%, it is considered effective. Follow up evaluations will be conducted on the 7th, 14th, 30th, 60th, 90th, and 180th day after intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided
Sharing research data requires hospital authorization and consent.

REFERENCES:
- [Result] Teo WP, Kannan A, Loh PK, Chew E, Sharma VK, Chan YC. Poor Tolerance of Motor Cortex rTMS in Chronic Migraine. J Clin Diagn Res. 2014 Sep;8(9):MM01-2. doi: 10.7860/JCDR/2014/9377.4886. Epub 2014 Sep 20. PMID 25386478
- [Result] Kalita J, Kumar S, Singh VK, Misra UK. A Randomized Controlled Trial of High Rate rTMS Versus rTMS and Amitriptyline in Chronic Migraine. Pain Physician. 2021 Sep;24(6):E733-E741. PMID 34554691